CLINICAL TRIAL: NCT06663930
Title: New Approach for Ovarian PRP Injection for Poor Responders ; Aiming At the Highest Response Rate
Brief Title: New Approach for Ovarian PRP Injection for Poor Responders
Status: Active, not recruiting | Type: Observational
Sponsor: Bassem Ayman Mahmoud Assaf (Other)
Responsible Party: Sponsor-Investigator, Bassem Ayman Mahmoud Assaf, Medical Doctor, Benha University
Organization: Benha University (Other)
Other Study IDs: New Approach For Ovarian PRP
Record Dates: First submitted 2024-10-19; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Poor Responders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

SUMMARY:
New Approach For Ovarian PRP Injection for poor responders

DETAILED DESCRIPTION:
Poor ovarian responders are at high risk of unsuccessful IVF/ICSI trials. In the last few years, many studies showed significant improvement of ovarian reserve parameters after PRP injection. There was no consensus regarding the route of injection, the volume injected, the location of PRP injection inside the ovary, the number of injection and the number of the cycle in which PRP is injected.

ELIGIBILITY:
Inclusion Criteria:

* AMH : < 0.5 ng/ml
* FSH: > 10 miu but < 25 miu.
* AFC : < 5 in both ovaries
* Poor ovarian response, in a previous IVF/ICSI trial , resulting in 3 or fewer oocytes.
* Normal uterine cavity , demonstrated by a recent hysteroscopy

Exclusion Criteria:

* Primary ovarian insufficiency with FSH > 25 miu.
* Previous ovarian surgery or Chemotherapy.
* On going Anticoagulant use.
* Carcinomas or a history of chronic pelvic pain.
* Present infection.
* Hemoglobin level lower than 11 g/L
* platelet count lower than 150 x 10³/μL.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: women attending their attempt of IVF/ICSI at Assaf Fertility center, after poor ovarian response in a previous trial, during the period March 2024 to June 2025
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PRP effect on ovary for better fertility outcome | one year
  This is a prospective cohort clinical observational study. Aiming at evaluating the clinical effects of injecting PRP(Platelet Rich Plasma) into ovaries, of poor responders, taking all measures which may improve the response rate. That is why we will inject PRP for 2 consecutive cycles, the first cycle via laparoscopy and the next cycle, via ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, benha, Egypt